CLINICAL TRIAL: NCT01137136
Title: Aromatase (CYP19) Polymorphism Between AI-responsive and AI-resistant Breast Cancer in Korea
Acronym: CYP19
Status: Suspended | Type: Observational
Why Stopped: Because of economic issue, we could just enrolled total 150 patients.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seok Jin Nam, Professor, M.D., Ph.D., Samsung Medical Center
Other Study IDs: 2009-11-035
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Polymorphism; CYP19; Aromatase Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SMAC (SMc AI user Cohort): All patients who took the AI (Aromatase inhibitor)will be enrolled

SUMMARY:
Aromatase(CYP19)inhibitor is one of the major antihormonal drug for breast cancer in postmenopausal women. The variation of CYP19 may affect the effect of aromatase inhibitor. However, the incidence of variation of CYP19 in Korea has not known. Therefore, the investigators want to know the incidence of variation of CYP19 and to assess the effect of these variations of CYP19 to aromatase inhibitor users.

ELIGIBILITY:
Inclusion Criteria:

* hormone receptor positiveBreast cancer patient
* postmenopausal women
* first user of aromatase inhibitor

Exclusion Criteria:

* premenopausal
* The patient who take the other antihormonal therapy
* osteoporosis patients

Max Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausa women who underwent surgery for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of CYP19 polymorphism | 12. 31. 2011

SECONDARY OUTCOMES:
The effect of CYP19 polymorphism to the prognosis of AI user | 12. 31. 2016

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Nam, M.D., Ph.D., Study Director — Samsung Medical Center, Sungkyunkwan University School of Medicine, Department of Surgery
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea